CLINICAL TRIAL: NCT07243236
Title: "Assessment of the Impact of Vaccine Funding by the National Health Insurance on Vaccination Coverage Among Patients Targeted by Current Vaccination Recommendations and Followed in Outpatient Consultations in Ile-de-France Region in France""
Brief Title: Impact of Vaccine Funding by the National Health Insurance on Vaccination Coverage Among Patients Targeted by Current Vaccination Recommendations and Followed in Outpatient Consultations
Acronym: VAXINOVA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence régionale de santé Ile de France (Unknown); Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251228; 2025-A01886-43 (Other: France : Ministry of Health)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthcare Providers; Postpartum
Keywords: Vaccine coverage; Vaccine funding within healthcare institutions; Outpatient consultations
MeSH Terms: interventions — Surveys and Questionnaires; Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women in the immediate postpartum period: Women in the immediate postpartum period (during their stay in the maternity ward) who have declared their pregnancy to the National Health Insurance, covered under maternity benefits up to the 12th day following delivery
  Interventions: Other: Questionnaires for patients
- Patients eligible for pneumococcal vaccination: Patients eligible for pneumococcal vaccination who benefit from long-term illness coverage (ALD), state medical aid (AME), or complementary universal health coverage C2S
  Interventions: Other: Questionnaires for patients
- Healthcare providers: Vaccinating healthcare providers + Other healthcare providers involved in the operational aspects of the project (excluding health data)
  Interventions: Other: Questionnaires for healthcare providers

INTERVENTIONS:
Other: Questionnaires for patients — Questionnaires for patients
  Groups: Patients eligible for pneumococcal vaccination; Women in the immediate postpartum period
Other: Questionnaires for healthcare providers — Questionnaires for healthcare providers
  Groups: Healthcare providers

SUMMARY:
The objective of our study is to evaluate the impact of vaccine funding for patients seen in outpatient consultations within four healthcare institutions in the Ile-de-France region in France, made possible through the establishment of a tripartite agreement between the hospital group, the Île-de-France Regional Health Agency (ARS IDF), and the Primary Health Insurance Fund (CPAM).

DETAILED DESCRIPTION:
The aim of this project is to highlight whether dedicated funding for vaccine procurement in healthcare institutions can generate both individual and collective benefits in terms of improved vaccination coverage among vulnerable patients at infectious risk.

Should the data analysis demonstrate a positive impact on vaccination coverage among patients who attended outpatient consultations in the participating institutions during the study period, it is planned to approach the Directorate General for Health with a view to generalizing such agreements between healthcare institutions and local health insurance organizations, thereby enabling reimbursement of vaccines included in the national immunization schedule administered within these institutions.

Primary objective: To assess the impact of National Health Insurance (NHI) funding for vaccines made available in outpatient consultations on pertussis vaccination coverage among pregnant women and pneumococcal vaccination coverage among eligible patients, in accordance with current French recommendations and fully covered by NHI, across four healthcare institutions in the Île-de-France region.

Secondary objectives:

To evaluate:

* The influence of socio-economic determinants on patients' vaccination coverage;
* Changes in the practices of hospital healthcare professionals in outpatient consultations regarding the monitoring of their patients' vaccination status;
* Changes in practices related to the documentation of patient vaccinations to facilitate communication between healthcare institutions and primary care practitioners through the use of existing digital tools (hospital software, electronic vaccination record (CVE) in MonEspaceSanté).

ELIGIBILITY:
Inclusion Criteria:

For patients:

1. For the assessment of pneumococcal coverage among patients eligible for this vaccination:

   * Individuals aged 18 years or older,
   * Individuals followed in outpatient consultations within a department and healthcare institution participating in the project;
   * Individuals eligible for pneumococcal vaccination against according to current French recommendations,
   * Individuals meeting the eligibility conditions and receiving care under long-term illness coverage (ALD) or benefiting from complementary universal health coverage (C2S) or state medical aid (AME).
2. For the assessment of pertussis vaccination among pregnant women:

   * Women aged 18 years or older,
   * Women who have had at least one follow-up outpatient consultation from 20 weeks of gestation in a maternity ward participating in the project,
   * Women in the immediate postpartum period (during their maternity stay) who have given birth to one or more live children and delivered after 36 weeks of gestation,
   * Women who have declared their pregnancy and are covered under maternity insurance (i.e., from the first day of the sixth month of pregnancy until the 12th day after delivery).

For healthcare professionals: all vaccinating healthcare providers working in a participating department or center.

Exclusion Criteria:

* Individuals seen in settings other than outpatient consultations (day hospital, week hospital, conventional hospitalization, International Vaccination Center).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During a follow-up hospital consultation, for patients eligible for pneumococcal vaccination or for postpartum women eligible for pertussis vaccination during pregnancy, the healthcare professional proposes and completes a questionnaire with the patient during the consultation.
Sampling Method: Non-Probability Sample
Enrollment: 2920 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of subjects vaccinated against pneumococcal infections | Month 3
  Variation in the number of subjects vaccinated against pneumococcal infections (eligible subjects according to current recommendations) before (according to the usual intra-hospital organization) and after the implementation of the National Health Insurance funding for vaccines made available during outpatient consultations for the target populations across four healthcare institutions in the Ile-de-France region
Number of subjects vaccinated against pneumococcal infections | Month 18
  Number of subjects vaccinated against pneumococcal infections (eligible subjects according to current recommendations), before (according to the usual intra-hospital organization) the implementation of the National Health Insurance funding for vaccines made available during outpatient consultations for the target populations
Number of subjects vaccinated against pertussis | Month 3
  Variation in the number of subjects vaccinated against pertussis during pregnancy, before (according to the usual intra-hospital organization) and after the implementation of the National Health Insurance funding for vaccines made available during outpatient consultations for the target populations
Number of subjects vaccinated against pertussis | Month 18
  Variation in the number of subjects vaccinated against pertussis during pregnancy, before (according to the usual intra-hospital organization) and after the implementation of the National Health Insurance funding for vaccines made available during outpatient consultations for the target populations

SECONDARY OUTCOMES:
Associated factors | Month 3
  Factors associated with pertussis vaccination among pregnant women and pneumococcal vaccination among eligible patients (including vaccination pathway, socio-demographic and socio-economic factors, category of healthcare providers involved in pregnancy follow-up, etc.),
Associated factors | Month 18
  Factors associated with pertussis vaccination among pregnant women and pneumococcal vaccination among eligible patients (including vaccination pathway, socio-demographic and socio-economic factors, category of healthcare providers involved in pregnancy follow-up, etc.),
Frequency with which vaccination providers offer vaccinations to eligible patients for these vaccinations | Month 3
  Frequency with which vaccination providers offer pertussis vaccination to pregnant women and pneumococcal vaccination to eligible patients for these vaccinations
Frequency with which vaccination providers offer vaccinations to eligible patients for these vaccinations | Month 18
  Frequency with which vaccination providers offer pertussis vaccination to pregnant women and pneumococcal vaccination to eligible patients for these vaccinations
Frequency with which vaccinating healthcare providers administer vaccinations to eligible patients for this vaccination | Month 3
  Frequency with which vaccinating healthcare providers administer pertussis vaccination to pregnant women and pneumococcal vaccination to eligible patients for this vaccination
Frequency with which vaccinating healthcare providers administer vaccinations to eligible patients for this vaccination | Month 18
  Frequency with which vaccinating healthcare providers administer pertussis vaccination to pregnant women and pneumococcal vaccination to eligible patients for this vaccination
Proportion of vaccinating healthcare providers | Month 3
  Proportion of vaccinating healthcare providers recording in a digital tool pertussis vaccinations for pregnant women and pneumococcal vaccinations for eligible patients
Proportion of vaccinating healthcare providers | Month 18
  Proportion of vaccinating healthcare providers recording in a digital tool pertussis vaccinations for pregnant women and pneumococcal vaccinations for eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Marie LACHATRE, MD, Study Director — Hôpital Cochin - APHP; Muriel BELIAH-NAPPEZ, MD, Study Chair — Agence régionale de santé Ile de France
Locations (6):
- France (6):
  - COCHIN HOSPITAL - Assistance Publique-Hôpitaux de Paris (APHP), Paris, IDF
  - Sud Seine Et Marne Hospital, Fontainebleau
  - Sud Seine Et Marne Hospital, Montereau-Fault-Yonne
  - Sud Seine Et Marne Hospital, Nemours
  - Rambouillet Hospital, Rambouillet
  - Delafontaine Hospital, Saint-Denis

REFERENCES:
- [Background] Chen H, Matsumoto H, Horita N, Hara Y, Kobayashi N, Kaneko T. Prognostic factors for mortality in invasive pneumococcal disease in adult: a system review and meta-analysis. Sci Rep. 2021 Jun 4;11(1):11865. doi: 10.1038/s41598-021-91234-y. PMID 34088948
- [Background] Schnell D, Mayaux J, de Bazelaire C, Legoff J, Feuillet S, Scieux C, Andreu-Gallien J, Darmon M, Baruchel A, Schlemmer B, Azoulay E. Risk factors for pneumonia in immunocompromised patients with influenza. Respir Med. 2010 Jul;104(7):1050-6. doi: 10.1016/j.rmed.2010.01.021. Epub 2010 Feb 24. PMID 20181467
- [Background] Belsky JA, Tullius BP, Lamb MG, Sayegh R, Stanek JR, Auletta JJ. COVID-19 in immunocompromised patients: A systematic review of cancer, hematopoietic cell and solid organ transplant patients. J Infect. 2021 Mar;82(3):329-338. doi: 10.1016/j.jinf.2021.01.022. Epub 2021 Feb 4. PMID 33549624
- [Background] Garcia Garrido HM, Knol MJ, Heijmans J, van Sorge NM, Sanders EAM, Klumpen HJ, Grobusch MP, Goorhuis A. Invasive pneumococcal disease among adults with hematological and solid organ malignancies: A population-based cohort study. Int J Infect Dis. 2021 May;106:237-245. doi: 10.1016/j.ijid.2021.03.072. Epub 2021 Mar 26. PMID 33781907
- [Background] Marijam A, Vroom N, Bhavsar A, Posiuniene I, Lecrenier N, Vroling H. Systematic Literature Review on the Incidence of Herpes Zoster in Populations at Increased Risk of Disease in the EU/EEA, Switzerland, and the UK. Infect Dis Ther. 2024 May;13(5):1083-1104. doi: 10.1007/s40121-024-00963-w. Epub 2024 Apr 24. PMID 38656653
- [Background] Ellington S, Strid P, Tong VT, Woodworth K, Galang RR, Zambrano LD, Nahabedian J, Anderson K, Gilboa SM. Characteristics of Women of Reproductive Age with Laboratory-Confirmed SARS-CoV-2 Infection by Pregnancy Status - United States, January 22-June 7, 2020. MMWR Morb Mortal Wkly Rep. 2020 Jun 26;69(25):769-775. doi: 10.15585/mmwr.mm6925a1. PMID 32584795
- [Background] Mertz D, Geraci J, Winkup J, Gessner BD, Ortiz JR, Loeb M. Pregnancy as a risk factor for severe outcomes from influenza virus infection: A systematic review and meta-analysis of observational studies. Vaccine. 2017 Jan 23;35(4):521-528. doi: 10.1016/j.vaccine.2016.12.012. Epub 2016 Dec 23. PMID 28024955
- [Background] Tubiana S, Belchior E, Guillot S, Guiso N, Levy-Bruhl D; Renacoq Participants. Monitoring the Impact of Vaccination on Pertussis in Infants Using an Active Hospital-based Pediatric Surveillance Network: Results from 17 Years' Experience, 1996-2012, France. Pediatr Infect Dis J. 2015 Aug;34(8):814-20. doi: 10.1097/INF.0000000000000739. PMID 25955837
- [Background] Fell DB, Johnson J, Mor Z, Katz MA, Skidmore B, Neuzil KM, Ortiz JR, Bhat N. Incidence of laboratory-confirmed influenza disease among infants under 6 months of age: a systematic review. BMJ Open. 2017 Sep 7;7(9):e016526. doi: 10.1136/bmjopen-2017-016526. PMID 28882916
- [Background] Del Riccio M, Spreeuwenberg P, Osei-Yeboah R, Johannesen CK, Fernandez LV, Teirlinck AC, Wang X, Heikkinen T, Bangert M, Caini S, Campbell H, Paget J; RESCEU Investigators. Burden of Respiratory Syncytial Virus in the European Union: estimation of RSV-associated hospitalizations in children under 5 years. J Infect Dis. 2023 Nov 28;228(11):1528-1538. doi: 10.1093/infdis/jiad188. PMID 37246724
- [Background] Wyplosz B, Fernandes J, Sultan A, Roche N, Roubille F, Loubet P, Fougere B, Moulin B, Duhot D, Vainchtock A, Raguideau F, Lortet-Tieulent J, Blanc E, Moisi J, Goussiaume G. Pneumococcal and influenza vaccination coverage among at-risk adults: A 5-year French national observational study. Vaccine. 2022 Aug 5;40(33):4911-4921. doi: 10.1016/j.vaccine.2022.06.071. Epub 2022 Jul 7. PMID 35811205
- [Background] Loubet P, Rouviere J, Merceron A, Launay O, Sotto A, On Behalf Of The Avnir Group. Patients' Perception and Knowledge about Influenza and Pneumococcal Vaccination during the COVID-19 Pandemic: An Online Survey in Patients at Risk of Infections. Vaccines (Basel). 2021 Nov 22;9(11):1372. doi: 10.3390/vaccines9111372. PMID 34835303
- [Background] Launay O, Le Strat Y, Tosini W, Kara L, Quelet S, Levy S, Danan J, Reveillon J, Houdayer J, Bouvet E, Levy-Bruhl D; ANRS-FORMVAC Study Group. Impact of free on-site vaccine and/or healthcare workers training on hepatitis B vaccination acceptability in high-risk subjects: a pre-post cluster randomized study. Clin Microbiol Infect. 2014 Oct;20(10):1033-9. doi: 10.1111/1469-0691.12689. Epub 2014 Jul 25. PMID 24850059
- [Background] Alessandrini V, Anselem O, Girault A, Mandelbrot L, Luton D, Launay O, Goffinet F. Does the availability of influenza vaccine at prenatal care visits and of immediate vaccination improve vaccination coverage of pregnant women? PLoS One. 2019 Aug 1;14(8):e0220705. doi: 10.1371/journal.pone.0220705. eCollection 2019. PMID 31369626
- [Background] Mohammed H, McMillan M, Roberts CT, Marshall HS. A systematic review of interventions to improve uptake of pertussis vaccination in pregnancy. PLoS One. 2019 Mar 28;14(3):e0214538. doi: 10.1371/journal.pone.0214538. eCollection 2019. PMID 30921421
- [Background] Du P, Jin S, Lu S, Wang L, Ma X, Wang J, Huang R, Luo Q, Yang S, Feng X. Strategies to increase the coverage of influenza and pneumonia vaccination in older adults: a systematic review and network meta-analysis. Age Ageing. 2024 Mar 1;53(3):afae035. doi: 10.1093/ageing/afae035. PMID 38476102